CLINICAL TRIAL: NCT04878367
Title: Behavioral Interventions to Reduce Particulate Matter Exposure in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021-0956
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: COPD without intervention group , with intervention group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD_E (Experimental): COPD patients with intervention
  Interventions: Behavioral: Five active practices of living rules for responding to fine dust.
- COPD_C (No Intervention): COPD patients without intervention

INTERVENTIONS:
Behavioral: Five active practices of living rules for responding to fine dust. — 1. Check the fine dust weather forecast
  2. Check the operation time and filter of the air purifier
  3. Window ventilation
  4. Inhalant is used or not
  5. Bad fine dust: Refrain from going out
  Arms: COPD_E

SUMMARY:
It is a prospective, multi-institutional clinical study and targets patients diagnosed with chronic obstructive pulmonary disease. About 120 subjects (35 at Ilsan Paik Hospital, 35 at Severance Hospital, and 50 at Asan Medical Center in Seoul) will be subject to a random allocation of 1:1. The arbitration group implements living rules for responding to fine dust, supports air purifiers, and only general guidance is implemented in the non-property group. Patients are recruited from Asan Medical Center in Seoul (Songpa-gu, Seoul), Severance Hospital ( Seodaemun-gu, Seoul), and Ilsan Paik Medical Center (Goyang, Gyeonggi-do) for 12 months. During outpatient visits, lung function tests and airway resistance tests shall be conducted, and surveys presented in the research plan shall be conducted.

DETAILED DESCRIPTION:
It is a prospective and multi-institutional clinical study targeting patients with chronic obstructive pulmonary disease in general.

A total of 120 COPD patients will be recruited from three institutions: Asan Medical Center, Severance Hospital, and Ilsan Paik Hospital. (60/30/30 expected) A panel of COPD patients is established to conduct prospective studies, and measures to mediate recurrence and deterioration of adult chronic respiratory diseases due to exposure to fine dust are presented. Improvement of the lifestyle of the arbitration forces. Detailed research methods such as air purifier support are presented in the research plan.

In addition, a fine dust measurement researcher visits each household to measure indoor fine dust concentration. The measurement method of fine dust concentration will be using the process test method, IoT-based sensors, and direct-to-read measuring devices to measure Air Korea's air pollution. Detailed visit timing and methods are carried out in the manner specified in the research plan.

We collect sputum at every visit and blood at the last visit.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Waste function test results show FEV1/FVC<0.7, FEV1 <80% of forecast

Exclusion Criteria:

* Patients under 18 years of age with changes in medication (such as inhalants).
* Older people over 80 years of age.
* People with no respiratory symptoms with mMRC 0.
* Who doesn't understand a simple explanation for fine dust exposure devices.
* Someone who disagrees with the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
SGRQ-C | 12 months
  Quality of life
CAT | 12 months
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sei won Lee, Principal Investigator — Seoul Asan Hospital
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The resident registration number may be used when requesting data from the National Statistical Office or the Health Review and Assessment Service for future research analysis and data collection.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data are available at the time of the analysis of the results after the clinical study.
Access Criteria: Gender, age, smoking power and address are collected anonymously.

REFERENCES:
- [Derived] Ji HW, Kang J, Kim HC, Jung J, Lee SJ, Jung JY, Lee SW. The association between cumulative exposure to PM2.5 and DNA methylation measured using methyl-capture sequencing among COPD patients. Respir Res. 2024 Sep 9;25(1):335. doi: 10.1186/s12931-024-02955-3. PMID 39251997
- [Derived] Kang J, Kim HC, Jang Y, Lee JB, Lee JS, Oh YM, Ji HW, Jung JY, Lee SW. Randomised controlled trial of a behavioural intervention to reduce exposure to PM2.5 in patients with COPD. Environ Int. 2023 Nov;181:108286. doi: 10.1016/j.envint.2023.108286. Epub 2023 Oct 24. PMID 37918066
- [Derived] Kang J, Jung JY, Huh JY, Ji HW, Kim HC, Lee SW. Behavioral interventions to reduce particulate matter exposure in patients with COPD. Medicine (Baltimore). 2021 Dec 10;100(49):e28119. doi: 10.1097/MD.0000000000028119. PMID 34889270